CLINICAL TRIAL: NCT04409639
Title: Phase 2 Trial of Cobimetinib in Newly Diagnosed or HMA-treated CMML Patients With RAS Pathway Mutations
Brief Title: Cobimetinib in Newly Diagnosed or HMA-treated CMML Patients With RAS Pathway Mutations
Acronym: CONCERTO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI132394
Record Dates: First submitted 2020-05-20; First posted 2020-06-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — cobimetinib

STUDY DESIGN:
Intervention Model Description: open-label, nonrandomized phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental): Cobimetinib is taken on a 28-day cycle. Each dose consists of three 20 mg tablets (60 mg) and should be taken once daily for 21 consecutive days (Days 1 to 21-treatment period); followed by a 7-day break (Days 22 to 28-treatment break). Each subsequent cobimetinib treatment cycle should start after a 7-day treatment break has elapsed.
  Interventions: Drug: Cobimetinib

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib is taken on a 28-day cycle. Each dose consists of three 20 mg tablets (60 mg) and should be taken once daily for 21 consecutive days (Days 1 to 21-treatment period); followed by a 7-day break (Days 22 to 28-treatment break). Each subsequent cobimetinib treatment cycle should start after a 7-day treatment break has elapsed.

SUMMARY:
This is an open-label, nonrandomized phase 2 trial to assess the efficacy of cobimetinib in RAS pathway activated CMML.

All eligible patients will be treated daily with cobimetinib in 28-day cycles. Cobimetinib will be administered for three weeks followed by a one week break prior to the start of the following cycle. Patients will remain on study therapy until treatment discontinuation criteria is met.

DETAILED DESCRIPTION:
This is an open-label, nonrandomized phase 2 trial to assess the efficacy of cobimetinib in RAS pathway activated CMML. Two cohorts of patients will be accrued using Simon's two-stage design (Simon, 1989) for both cohorts. Cohort 1 will enroll nine newly diagnosed patients in the first stage and if four or more responses are observed five additional patients will be enrolled in the second stage. Cohort 2 will enroll six HMA refractory patients in the first stage and if one or more responses are observed then nine additional patients will be enrolled in the second stage.

All eligible patients will be treated daily with cobimetinib in 28-day cycles. Cobimetinib will be administered consecutively for three weeks followed by a one week break prior to the start of the following cycle. Patients will remain on study therapy until treatment discontinuation criteria is met.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Newly diagnosed or hypomethylating agent (HMA) refractory chronic myelomonocytic leukemia (CMML -0/-1/-2; 2016 WHO classification) with RAS pathway activation as determined by standard of care hematopoietic cell sequencing results on peripheral blood or bone marrow demonstrating NRAS, KRAS, PTPN11, FLT3, CBL, JAK2, BRAF or NF1 mutations at variant allele frequency ≥ 5%. BMBx, NGS, FISH or BCR-ABL1 PCR, and cytogenetics should be done at the primary trial site within 21 days prior to C1D1. 5.1.2 If the patient is FLT3-ITD positive, the FLT3-ITD PCR allelic ratio must be ≥ 0.05 on testing done on screening biopsy (NOTE: cannot quantitate FLT3-ITD VAF by NGS, must be a separate PCR test).
* ECOG Performance Status ≤ 3.
* Adequate organ function as defined as:

  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * Unless elevation is related to Gilbert's syndrome, hemolysis, or thought to be due to leukemic hepatic involvement.
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN ----Unless elevation is related to leukemic hepatic involvement.
  * Renal:

    ---Serum creatinine ≤ 2x ULN
  * OR

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:
    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
    * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
* Left ventricular function ≥ 50% as assessed by echocardiogram.
* Negative pregnancy test for women of childbearing potential or evidence of post-menopausal status. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Highly effective contraception for both male and female subjects throughout the study and at least 3 months after the last dose of study therapy as described in Section 7.4 of the protocol.
* Recovery to baseline or Grade ≤ 1 CTCAE v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Previous exposure to experimental MEK inhibitors for CMML.
* Grade 2 or greater QTc prolongation on screening electrocardiogram (ECG) or clinically significant cardiovascular disease (uncontrolled or symptomatic atrial arrhythmias, congestive heart failure, myocardial infarction/CABG/PCI within 6 months of screening, uncontrolled arterial hypertension or history of ventricular arrhythmia)
* Clinical or laboratory evidence of central nervous system (CNS) leukemia.
* Major surgery within 4 weeks prior to study drug initiation.
* History of interstitial lung disease.
* History of retinal detachment, central serous retinopathy (CSR), retinal vein occlusion (RVO), or at high risk for CSR or RVO following screening ophthalmologic exam at discretion of PI/Sub-I following review of exam findings, and, if necessary, consultation with ophthalmology provider.
* Patients with muscular and/or neuromuscular disorders associated with elevated CPK (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, or spinal muscular atrophy).
* Any active significant gastrointestinal dysfunction as determined by the clinical investigator to interfere with the patient's ability to swallow or absorb the study treatment, (i.e. refractory nausea and vomiting, malabsorption and external biliary shunt).
* Pregnant or nursing (lactating) women.
* On chronic treatment with strong CYP3A inhibitors or patients taking St. John's Wort, carbamazepine, efavirenz, phenytoin, rifampin, and other strong and moderate CYP3A inducers.
* Diagnosis of any other malignancy within 2 years before study enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or cervix, low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (eg, surgery, radiation, or castration), or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms, or any solid tumor malignancy that has been adequately treated for which there is no evidence of disease. Patients with monoclonal gammopathy of undetermined significance (MGUS) are permitted to enroll.
* Known HIV infection with a detectable viral load at the time of screening.

  --Note: Patients on effective antiretroviral therapy with an undetectable viral load at the time of screening are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Subjects taking prohibited medications as described in Section 6.3.2. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur before the start of treatment.
* Known prior severe hypersensitivity to cobimetinib or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate defined as the proportion of patients achieving complete remission, complete cytogenetic remission, partial remission, marrow response, and clinical benefit according to the 2015 MDS/MPN-IWG criteria | From 1st dose of study medication to decision to end treatment or up to 12 months of treatment, whichever came first
  assess the efficacy of cobimetinib in patients with newly diagnosed and HMA- refractory chronic myelomonocytic leukemia (CMML)

SECONDARY OUTCOMES:
Frequency of adverse events characterized by seriousness, severity (CTCAEv5.0), duration and relationship to study therapy. | Until decision to end treatment or up to 12 months of treatment, whichever came first
  assess the safety of cobimetinib treatment in CMML
Proportion of patients achieving complete response complete response (CR) + partial response (PR) | Until decision to end treatment or up to 12 months of treatment, whichever came first
  Assessment of complete response (CR) + partial response (PR) rate (defined by 2015 MDS/MPN-IWG criteria)
Progression-free survival (PFS) | up to 36 months after the start of therapy, the time of progression, initiation of alternative treatment or death, whichever came first
  Assessment of long-term efficacy
Overall Survival (OS) | Study anticipated to be 60 months.
  Assessment of long-term efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Ami Patel, MD, Principal Investigator — Huntsman Cancer Institute
Locations (3):
- United States (3):
  - Oregon Health and Science University, Portland, Oregon
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No